CLINICAL TRIAL: NCT00361257
Title: Phase II, Randomized, Placebo-Controlled, Double-Blind Study of Minocycline in the Treatment of HIV-Associated Cognitive Impairment
Brief Title: Minocycline for the Treatment of Decreased Mental Function in HIV-Infected Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated early due to futility.
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Neurologic AIDS Research Consortium (NARC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG A5235; 1U01AI068636 (NIH)
Record Dates: First submitted 2006-08-04; First posted 2006-08-08 (Estimated); Results first posted 2011-07-26 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Minocycline; Tetracycline

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Minocycline (Experimental): 100 mg orally every 12 hours
  Interventions: Drug: Minocycline
- Arm 2: Matching placebo (Placebo Comparator): orally every 12 hours
  Interventions: Drug: Placebo (Tetracycline)

INTERVENTIONS:
Drug: Minocycline — Tetracycline antibiotic, 100 mg taken orally every 12 hours
  Arms: Arm 1: Minocycline
Drug: Placebo (Tetracycline) — Tetracycline antibiotic placebo, orally every 12 hours
  Arms: Arm 2: Matching placebo

SUMMARY:
The purpose of this study is to determine the effectiveness of minocycline, an antibiotic, in lessening the decreased mental function sometimes caused by anti-HIV drugs.

DETAILED DESCRIPTION:
Cognitive impairment, including disabling cognitive, behavioral, and social dysfunction, continues to be a major problem faced by HIV-infected people taking antiretroviral therapy (ART). Research is needed to develop treatment that can be given alongside ART to prevent or lessen cognitive impairment caused by ART. Minocycline, an antibiotic commonly used for the treatment of acne and rheumatoid arthritis, has demonstrated anti-inflammatory and neuroprotective properties in previous studies. This study will evaluate the effectiveness of 24-week therapy with minocycline in lessening the cognitive impairment of HIV infected adults taking ART.

This study will last at least 24 weeks and has two steps. Patients will be stratified by HIV viral load and their neurocognitive state at study screening. In Step I, patients will be randomly assigned to one of two groups. Group 1 participants will receive twice-daily minocycline for 24 weeks; Group 2 participants will receive placebo. At the end of Phase I, study participants will be offered to enter Step II; all participants in Step II will receive twice-daily minocycline for an additional 24 weeks.

There will be a total of 8 study visits: 5 visits for Step I (including the entry visit) and 3 visits for Step II. Medical history will occur at all visits. Blood collection will occur at all visits. Participants who have positive nonreactive rapid plasma regain (RPR) values at screening will have mandatory lumbar punctures; for those with negative serum RPR results lumbar punctures are optional. Participants who test positive for syphilis will also have a lumbar puncture at their discretion to determine if syphilis has affected the brain. A neurological exam, other neuropsychological, dementia, and depression scale assessments, and urine collection will occur at most visits. Patients will be asked to complete a questionnaire on daily living at study entry and Weeks 12 and 24. Patients who have a lumbar puncture at Week 24 will receive a phone call 2 to 5 days after the procedure to report any adverse effects. Some participants may also have an electrocardiogram (ECG) during the study. For participants not on atazanavir some procedures and sample collections are optional.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Currently on a stable ART regimen for at least 16 consecutive weeks prior to study entry. Participants whose regimens have changed with respect to dose or formulation are eligible, but patients who have changed to different drugs in the same class are not eligible. Participants taking atazanavir must also be taking ritonavir or a ritonavir-boosted drug to be eligible for this study. More information on this criterion can be found in the protocol.
* Plan to stay on current ART regimen between study screening and Week 24
* AIDS Dementia Scale (ADC) Stage greater than 0
* Cognitive impairment, as evidenced by neuropsychological tests administered at screening
* Progressive neurocognitive decline. More information on this criterion can be found in the protocol.
* Estimated premorbid IQ of 70 or higher indicated by an age-corrected scaled score of 5 or higher on the vocabulary section of the Wechsler Adult Intelligence Scale Revised (WAIS-R) administered at study screening
* Karnofsky performance score of 60 or higher
* Ability to sit and stand for at least 2 hours and swallow medications with an 8-ounce glass of water
* Willing to use acceptable methods of contraception
* Willing to adhere to study schedule

Exclusion Criteria:

* Current cancers. Patients with basal cell carcinoma, in situ carcinoma of the cervix, or Kaposi's sarcoma without evidence of visceral involvement or cancer not requiring systemic chemotherapy are not excluded.
* Severe premorbid psychiatric illness, including schizophrenia and major depression, which, in the opinion of the investigator, may interfere with the study
* Active symptomatic AIDS-defining opportunistic infection within 45 days prior to study entry
* Previous or current confounding neurological disorders. More information on this criterion can be found in the protocol.
* Central nervous system infections or cancers. More information on this criterion can be found in the protocol.
* Systemic lupus
* Thyroid disease diagnosed within 24 weeks of study entry
* Active drug or alcohol abuse that, in the opinion of the investigator, may interfere with the study
* Serious illness requiring systemic treatment or hospitalization. Patients who complete therapy or are clinically stable on therapy are not excluded.
* Investigational agents within 45 days prior to study entry. Patients taking expanded access drugs or drugs used in an ACTG protocol for HIV treatment or for HIV-associated complications that are not prohibited by this protocol are not excluded.
* History of allergy/sensitivity to minocycline or other tetracyclines and their formulations
* Any esophageal or other condition that would interfere with a patient's ability to swallow study medication
* Participation in a previous clinical drug research trial of HIV-associated cognitive impairment. Patients who have had an objective decline in performance as defined by the protocol are not excluded.
* Any other clinically significant condition or laboratory abnormality that, in the opinion of the investigator, would interfere with the study
* Certain medications
* Certain abnormal laboratory values. Patients who test positive on nonreactive rapid plasma reagin tests (RPR)are not excluded.
* Inability to undergo lumbar punctures
* Breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2007-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ned Sacktor, MD, Study Chair — Department of Neurology, Johns Hopkins Bayview Medical Center
Locations (16):
- United States (16):
  - UCLA-David Geffen School of Medicine, Los Angeles, California
  - University of California, San Diego, California
  - University of Colorado Health Science Center, Denver, Colorado
  - The Ponce de Leon Ctr. CRS, Atlanta, Georgia
  - Northwestern University CRS, Chicago, Illinois
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Division of Infectious Diseases, Boston, Massachusetts
  - Henry Ford Hosp. CRS, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - NYU Med Ctr, Dept of Medicine, New York, New York
  - 1101 University of Rochester Medical Center, Division of Infectious Diseases, Rochester, New York
  - University of North Carolina, AIDS Clinical Trials Unit, Chapel Hill, North Carolina
  - The Research and Education Group - Portland CRS, Portland, Oregon
  - University of Pennsylvania, ACTU, Philadelphia, Pennsylvania
  - Virginia Commonwealth Univ. Medical Ctr. CRS, Richmond, Virginia
  - Univ of Washington, Harborview Medical Ctr, Seattle, Washington

REFERENCES:
- [Background] Bell JE. An update on the neuropathology of HIV in the HAART era. Histopathology. 2004 Dec;45(6):549-59. doi: 10.1111/j.1365-2559.2004.02004.x. PMID 15569045
- [Background] Ferrari S, Vento S, Monaco S, Cavallaro T, Cainelli F, Rizzuto N, Temesgen Z. Human immunodeficiency virus-associated peripheral neuropathies. Mayo Clin Proc. 2006 Feb;81(2):213-9. doi: 10.4065/81.2.213. PMID 16471077
- [Background] Zink MC, Uhrlaub J, DeWitt J, Voelker T, Bullock B, Mankowski J, Tarwater P, Clements J, Barber S. Neuroprotective and anti-human immunodeficiency virus activity of minocycline. JAMA. 2005 Apr 27;293(16):2003-11. doi: 10.1001/jama.293.16.2003. PMID 15855434
- [Result] Sacktor N, Miyahara S, Deng L, Evans S, Schifitto G, Cohen BA, Paul R, Robertson K, Jarocki B, Scarsi K, Coombs RW, Zink MC, Nath A, Smith E, Ellis RJ, Singer E, Weihe J, McCarthy S, Hosey L, Clifford DB; ACTG A5235 team. Minocycline treatment for HIV-associated cognitive impairment: results from a randomized trial. Neurology. 2011 Sep 20;77(12):1135-42. doi: 10.1212/WNL.0b013e31822f0412. Epub 2011 Sep 7. PMID 21900636
- [Result] Sacktor N, Miyahara S, Evans S, Schifitto G, Cohen B, Haughey N, Drewes JL, Graham D, Zink MC, Anderson C, Nath A, Pardo CA, McCarthy S, Hosey L, Clifford D; ACTG A5235 team. Impact of minocycline on cerebrospinal fluid markers of oxidative stress, neuronal injury, and inflammation in HIV-seropositive individuals with cognitive impairment. J Neurovirol. 2014 Dec;20(6):620-6. doi: 10.1007/s13365-014-0292-0. Epub 2014 Nov 7. PMID 25377444

RESULTS

PARTICIPANT FLOW:
Groups:
- Minocycline: 100 mg orally every 12 hours
- Matching Placebo: Placebo taken orally every 12 hours
Period: Step 1: Minocycline vs. Placebo
Arm/Group | Minocycline | Matching Placebo
Started | 52 | 55
Completed | 40 | 43
Not Completed | 12 | 12
Period: Step 2: Minocycline(Open Label) for All
Arm/Group | Minocycline | Matching Placebo
Started | 28 (40 participants completed Step 1; however,12 decided not to enroll Step 2,so 40-12=28 started Step 2) | 34 (43 participants completed Step 1; however, 9 decided not to enroll Step 2,so 43-9=34 started Step 2.)
Completed | 13 | 19
Not Completed | 15 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minocycline | Matching Placebo | Total
Number analyzed (Participants) | 52 | 55 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 54 | 106
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (7) | 52 (7) | 51 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 13 | 18
  Male | 47 | 42 | 89
Cognitive Performance Score NPZ-8 [Mean (Standard Deviation); unit: z-score] — Cognitive performance is measured by NPZ-8. The NPZ-8 is defined as the average of age and education adjusted z-scores of eight neuropsychological tests subcomponents in the neuropsychological test battery:
  1. Grooved Pegboard Dominant Hand (GPD)
  2. Grooved Pegboard Non-dominant hand (GPN)
  3. Choice Reaction Time (CRT)
  4. Sequential Reaction Time (QRT)
  5. Timed Gait (TIG)
  6. Trail Making Part A (TMA)
  7. Trail Making Part B (TMB)
  8. Symbol Digit (SYD)
  z-score | -0.75 (0.90) | -1.03 (0.98) | -0.90 (0.95)
Global Deficit Z-Score (GDS) [Mean (Standard Deviation); unit: z-score] — GDS is defined as the average of age and education adjusted z-scores of 14 individual deficit scores in the test battery, including Time Gait, Grooved Pegboard Test for the dominant and non-dominant hands, Trail Making Test parts A and B, Symbol Digit Test, simple and sequential reaction time - CalCAP, Hopkins Verbal Learning Test (Revised)- Learning, Delayed Recall and Recognition trials, and Stroop Color Interference Test-color, word, and interference tasks.
  z-score | -0.86 (0.72) | -1.08 (0.90) | -0.97 (0.82)
Cognitive Gross Motor Function Domain Z-Score [Mean (Standard Deviation); unit: z-score] — The cognitive gross motor function is age and education adjusted z-score of Timed Gait.
  z-score | -2.44 (3.10) | -3.66 (4.16) | -3.06 (3.71)
Fine Motor Function Domain Z-Score [Mean (Standard Deviation); unit: z-score] — This is an average z-scores of Grooved Pegboard Dominant and Non-Dominant Hand Tests adjusted for age, sex, education, and African-American ethnicity. The grooved pegboard is a manipulative dexterity test requiring rapid visual-motor coordination. The test is completed using the dominant hand (GPD) and then using the non-dominant hand (GPN). The score for each hand is the time in seconds that the participant takes to complete the entire board.
  z-score | -0.35 (0.96) | -0.73 (0.99) | -0.55 (0.99)
Psychomotor Function Domain Z-Score [Mean (Standard Deviation); unit: z-score] — This is an average of z-scores of Trail Making Part A (TMA) and Trail Making Part B (TMB) tests adjusted for age, sex, education, and African-American ethnicity. The TMA and TMB tests are measures of planning ability, visual-motor speed and concentration. Subjects are required to connect randomly placed numbers in sequence (1-25 for TMA) or to sequentially connect both numbers and letters while alternating back and forth (1-A-2-B-3-C-4-D etc. for TMB). Scores are the time in seconds required to complete the tasks.
  z-score | 0.15 (1.00) | 0.04 (1.03) | 0.10 (1.01)
Fine Motor/Nonverbal Function Domain Z-Score [Mean (Standard Deviation); unit: z-score] — This score is a age and education adjusted z score of Symbol Digit Test (SYD). This test assesses the participant's ability to maintain rapid visual-motor sequencing in a timed test. The score is the total number of correctly transcribed numbers in the time limit (90 seconds). Participants receive 1 point for each item filled in correctly.
  z-score | -1.11 (1.15) | -1.24 (1.18) | -1.18 (1.16)
Information Processing Function Domain Z-Score [Mean (Standard Deviation); unit: z-score] — This is the average age and education adjusted z-scores of simple and sequential reaction time tests adjusted for age and education.
  z-score | -1.05 (1.52) | -1.03 (1.49) | -1.04 (1.50)
Verbal Memory Domain Z-Score [Mean (Standard Deviation); unit: z-score] — This is the average of z-scores of Hopkins Verbal Learning Test- Revised, Learning and Delayed Recall Tests adjusted for age and education. The recognition test list comprises 24 words, consisting of 12 words from the original list and 12 "distracters". The subject must answer "yes" if the word was from the list and "no" otherwise. Twenty minutes after the third list from verbal learning and immediate recall, delayed recall is assessed by asking the subject to recall as many words as possible from the list. The score is the number of words that are correctly recalled from the original list.
  z-score | -1.33 (1.16) | -1.41 (1.12) | -1.37 (1.14)
Frontal Systems Function Domain Z-Score [Mean (Standard Deviation); unit: z-score] — This is the average age and education adjusted z-scores of Stroop Color Interference Test (CTP) and interference task (STP). The Stroop Task is a measure of divided attentional abilities. Performance is measured by the amount of time required to read each of three cards: (1) blocks of colors, (2) names of colors, and (3) colored words. For each task, the time (in seconds) is the score that should be recorded on the form. A task that cannot be completed in 240 seconds is scored as incomplete.
  z-score | -0.79 (0.98) | -1.05 (1.57) | -0.92 (1.32)
Karnofsky Score [Number; unit: participants] — Karnofsky performance score is ranged from 100 to 0:
  100: Normal; 90: Able to Carry on normal Activity; 80: Normal Activity with Effort; Some Signs or Symptoms of Disease; 70: Cares for Self, Unable to Carry on Normal Activity or to Do Active Work; 60: Requires Occasional Assistance but is Able to Care for Most of Needs; 50: Requires Considerable Assistance and Frequent Medical Care; 40: Disabled, Requires Special Care and Assistance; 30: Severely Disabled; Hospitalization Indicated Although Death is Not Imminent; 20: Very Sick; 10: Morbibund, Fatal Processes Progressing Rapidly; 0: Death
  participants
    70 | 5 | 0 | 5
    80 | 13 | 16 | 29
    90 | 21 | 34 | 55
    100 | 8 | 5 | 13
    missing | 5 | 0 | 5
Cluster of Differentiation 4 (CD4) [Mean (Standard Deviation); unit: copies/mm^3] — CD4 counts by group at baseline
  copies/mm^3 | 551.65 (312.96) | 535.49 (253.11) | 543.35 (282.53)
Cluster of Differentiation 8 (CD8) [Mean (Standard Deviation); unit: copies/mm^3] — CD8 counts by group at baseline
  copies/mm^3 | 925.58 (370.48) | 838.78 (353.73) | 880.96 (362.88)
HIV-1 Plasma RiboNucleic Acid (RNA) Viral Loads [Number; unit: participants] — HIV Plasma RNA viral load less than 30 copies/mL is undetectable, the values will be imputed as 30 copies/mL.
  participants
    Plasma RNA VL >=30 copies/mL | 7 | 6 | 13
    Plasma RNA VL < 30 copies/mL | 42 | 41 | 83
    missing | 3 | 8 | 11
HIV-1 CerebroSpinal Fluid (CSF) RNA Viral Loads (VL) [Number; unit: participants] — HIV CSF RNA viral load less than 30 copies/mL is undetectable, the values will be imputed as 30 copies/mL.
  participants
    CSF RNA VL >=30 copies/mL | 1 | 2 | 3
    CSF RNA VL <30 copies/mL | 20 | 18 | 38
    missing | 31 | 35 | 66
Central Nervous System (CNS) Penetration Score [Mean (Standard Deviation); unit: Scores on a scale] — The baseline CNS penetration score is calculated based on the revised CNS penetration-effectiveness ranks (provided by Dr. Scott Letendre). The score is simply a sum of the ranks of all drugs which participants took at baseline. The better the drug penetrates, the higher the score. The range of ranks are 1 to 4, so the CNS penetration score is integer numbers greater than 1.
  Scores on a scale | 7 (3) | 7 (3) | 7 (3)
Stratification Variable 1 - CSF Viral Load (VL) - Pre-baseline [Number; unit: participants] — Participants were stratified based on two factors. One is CSF HIV-1 RNA. This variable has three levels using the TaqMan assay in CSF: (1) HIV CSF RNA VLs ≥30 copies/mL (detectable), <30 copies/mL (Undetectable), or no lumbar punctures (LPs). The assessment was conducted BEFORE the baseline in order to use this information for randomization.
  participants
    CSF RNA VL < 30 copies/mL | 21 | 22 | 43
    CSF RNA VL >= 30 copies/mL | 3 | 4 | 7
    No Lumbar Punctures (LPs) | 28 | 29 | 57
Stratification Variable 2 - Objective or subjective Neuropsychological test - Pre-baseline [Number; unit: participants] — The 2nd stratification factor is progressive neurocognitive decline defined by objective or subjective criteria at pre-baseline. A decline of at least 1.0 standard deviation below age-matched and education-matched controls on two or more independent tests or 2.0 standard deviations below age-matched and education-matched controls on one test within 1 year before entry is defined as objective decline. Otherwise, subjective neurocognitive decline is defined by the participant or family member or caregiver AND a Center for Epidemiological Studies Depression score <16 within 45 days before entry.
  participants
    Objective Neuropsychological (NP) Test | 5 | 7 | 12
    Subjective NP Test | 47 | 48 | 95
Instrumental Activities of Daily Living (IADL) Summary Score [Mean (Standard Deviation); unit: Scores on a scale] — The IADL questionnaire has 16 common tasks: 1. Housekeeping; 2.Managing Finances; 3. Buying Groceries; 4.Cooking; 5. Planning Social Activities; 6.Understanding Reading Materials/TV; 7.Transportation; 8.Using the Telephone; 9.Home Repairs; 10.Bathing; 11.Dressing; 12.Shopping; 13.Laundry; 14.Taking/Keeping Track of Medication; 15.Child Care; 16.Work. For each task, if the score at the time of evaluation is worse than the best in the past, an indicator of 1 is given; otherwise 0. The IADL score is a sum of 16 indicators divided by 16. The lower score indicates better. The range is from 0 to 1.
  Scores on a scale | 0.12 (0.15) | 0.13 (0.16) | 0.12 (0.15)
Medication Management Test (MMT) Score [Mean (Standard Deviation); unit: Scores on a scale] — The medication management test (modified) is designed to assess participants' medication management ability and their own medications and management. It's the number of how many times participants correctly answered 16 questions.
  Scores on a scale | 14.72 (1.41) | 14.09 (2.52) | 14.39 (2.08)
Alternate Psychomotor Function Z-Score [Mean (Standard Deviation); unit: z-score] — This is the average of z scores of Trail Making Part A and Symbol Digit Tests. Trail Making Part A z score was adjusted for age, sex, education, and African-Ametrican ethnicity. Symbol Digit z score was adjusted for age and education.
  z-score | -0.54 (0.82) | -0.63 (0.92) | -0.58 (0.87)
Alternate Verbal Memory Z-Score [Mean (Standard Deviation); unit: z-score] — This is the average of age and education adjusted z scores of standardized trials 1 to 3 and delayed recall tests.
  z-score | -1.33 (1.16) | -1.41 (1.12) | -1.37 (1.14)
Alternate Frontal Systems Z-Score [Mean (Standard Deviation); unit: z-score] — This is average of z scores of standardized interference task and trailmaking part b tests. The interference task z score was adjusted for age and education. The trailmaking part b z score was adjusted for age, sex, education, and African-American ethnicity.
  z-score | -0.04 (0.86) | -0.13 (1.09) | -0.09 (0.98)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Performance Compared to Baseline
Description: Th cognitive performance is measured by NPZ-8. NPZ-8 is defined as the average of age and education adjusted z-scores of eight neuropsychological tests subcomponents in the neuropsychological test battery. These eight tests are:
  1. Grooved Pegboard Dominant Hand (GPD)
  2. Grooved Pegboard Non-dominant hand (GPN)
  3. Choice Reaction Time (CRT)
  4. Sequential Reaction Time (QRT)
  5. Timed Gait (TIG)
  6. Trail Making Part A (TMA)
  7. Trail Making Part B (TMB)
  8. Symbol Digit (SYD) The primary outcome is NPZ-8 score at week24 - NPZ-8 score at baseline.
Time Frame: At baseline and week 24
Population: The descriptive statistics above were based on the observed data; however, the statistical analysis was conducted by the ITT analysis and the missing outcomes at week 24 were imputed based on multiple regression imputations.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 41 | 48
z-score | 0.12 (0.71) | 0.17 (0.67)
Statistical Analysis 1: Comparison: Minocycline vs Matching Placebo; The null hypothesis was that the 24-week change of NPZ-8 in the minocycline group was the same as the one in the placebo group; Test type: Superiority or Other; p = 0.651, Regression, Linear — The p-value was not adjusted for multiple comparisons; The model was adjusted for stratification variables, the CNS penetration score, and the baseline NPZ-8 score; Slope = 0.064, 95% CI 2-sided [-0.258 to 0.386], Standard Error of Mean 0.164 — The total number used for the statistical analysis was 107 (52 in the minocycline arm and 55 in the placebo arm)

2. Secondary Outcome: Change in Global Deficit Z-Score (GDS)
Description: GDS on the test battery is the simple average of all 14 individual deficit scores in the test battery, including Time Gait, Grooved Pegboard Test for the dominant and non-dominant hands, Trail Making Test parts A and B, Symbol Digit Test, simple and sequential reaction time - CalCAP, Hopkins Verbal Learning Test (Revised)- Learning, Delayed Recall and Recognition trials, and Stroop Color Interference Test-color, word, and interference tasks. The outcome is the 24 week change of GDS Z-score (24 week-baseline).
Time Frame: At baseline and week 24
Population: The analysis was based on the observed data.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 41 | 48
z-score | 0.11 (0.58) | 0.09 (0.51)
Statistical Analysis 1: Comparison: Minocycline vs Matching Placebo; The null hypothesis was that the 24-week changes in Global Deficit Score (GDS) between the minocycline and placebo groups are the same; Test type: Superiority or Other; p = 0.434, Regression, Linear — The p-value was not adjusted for multiple comparisons; The model was adjusted for stratification variables, the CNS penetration score, and the baseline GDS score; Slope = 0.091, 95% CI 2-sided [-0.140 to 0.323], Standard Error of Mean 0.116

3. Secondary Outcome: Change in Investigator's Clinical Global Impression Score (ICGIS)
Description: Clinicians were asked to rate their overall impression about the clinical improvement or worsening of his/her study participants. They can choose from the following 7 levels: (0) No Change, (1) Mild Improvement, (2) Moderate Improvement, (3) Marked Improvement, (4) Mild Worsening, (5) Moderate Worsening, and (6) Marked Worsening.
  For the analysis, we simplified the outcome into the following 3 levels: (0) worsened, (1) No Change, and (2) Improved.
Time Frame: At week 24
Population: The analysis was based on observed data.
Measure: Number; unit: participants
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 41 | 45
participants
  Worsened | 4 | 2
  No Change | 28 | 31
  Improved | 9 | 12
Statistical Analysis 1: Comparison: Minocycline vs Matching Placebo; The null hypothesis is that the 24 week changes of participants' clinical status in the minocycline group were the same as the ones in the placebo group based on ICGIS; Test type: Superiority or Other; p = 0.337, Regression, Cumulative Logistic — The p-value was not adjusted for multiple comparisons; The model was adjusted for the stratification variables and the CNS penetration score; Odds Ratio (OR) = 1.569, 95% CI 2-sided [0.625 to 3.936], Standard Deviation 0.469

4. Secondary Outcome: Change in Cognitive Gross Motor Function Domain Z-Score
Description: The cognitive gross motor function is a age and education adjusted z score of Timed Gait (TIG). The outcome is the 24 week change of cognitive gross motor function domain z-scores (week 24-baseline).
Time Frame: At baseline and week 24
Population: The analysis was based on the observed data.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 41 | 42
z-score | 0.22 (1.61) | 0.08 (2.68)
Statistical Analysis 1: Comparison: Minocycline vs Matching Placebo; The null hypothesis is that the 24 week change in the cognitive gross motor function domain score in the minocycline group is the same as the one in the placebo group; Test type: Superiority or Other; p = 0.243, Regression, Linear — The p-value was not adjusted for multiple comparisons; The model was adjusted for the stratification variables, the CNS penetration score, and the baseline cognitive gross motor function domain score; Slope = 0.502, 95% CI 2-sided [-0.349 to 1.354], Standard Error of Mean 0.428

5. Secondary Outcome: Change in Fine Motor Function Domain Z-Score
Description: The fine motor function domain score is an average of age, sex, education, and African-American ethnicity adjusted z scores of Grooved Pegboard Dominant Hand (GPD) and Grooved Pegboard Non-dominant hand (GPN). The outcome is a 24 week change of the fine motor function domain z-score (week 24-baseline).
Time Frame: At baseline and week 24
Population: The analysis was based on observed data.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 41 | 48
z-score | 0.27 (0.84) | 0.05 (0.61)
Statistical Analysis 1: Comparison: Minocycline vs Matching Placebo; The null hypothesis was that the 24 week change in fine motor function domain score in the minocycline group was the same as the one in the placebo group; Test type: Superiority or Other; p = 0.059, Regression, Linear — The p-value was not adjusted for multiple comparisons; The model was adjusted for the stratification variables, the CNS penetration score, and the baseline fine motor function domain score; Slope = 0.293, 95% CI 2-sided [-0.011 to 0.596], Standard Error of Mean 0.153

6. Secondary Outcome: Change in Psychomotor Function Domain Z-Score
Description: The psychomotor function domain score us the average of age, sex, education, and African-American ethnicity adjusted z scores of Trail Making Part A (TMA) and Trail Making Part B (TMB). The outcome is the 24 week change of psychomotor function domain z-scores (week24-baseline).
Time Frame: At baseline and week 24
Population: The analysis was based on observed data.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 41 | 48
z-score | 0.07 (0.66) | 0.15 (0.88)
Statistical Analysis 1: Comparison: Minocycline vs Matching Placebo; The null hypothesis was that the 24 change of psychomotor function domain score in the minocycline group is the same as in the placebo group; Test type: Superiority or Other; p = 0.572, Regression, Linear — The p-value was not adjusted for multiple comparisons; The model was adjusted for stratified variables, the baseline CNS penetration score, and the baseline psychomotor function domain score; Slope = -0.083, 95% CI 2-sided [-0.375 to 0.209], Standard Error of Mean 0.147

7. Secondary Outcome: Change in Fine Motor/Nonverbal Function Domain Z-Score
Description: The fine motor/nonverbal function domain score is a age and education adjusted z score of Symbol Digit Test (SYD) The outcome is the 24 change of fine motor/nonverbal function domain z-score (week 24-baseline).
Time Frame: At baseline and week 24
Population: The analysis was based on observed data.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 41 | 48
z-score | -0.15 (0.76) | -0.07 (0.92)
Statistical Analysis 1: Comparison: Minocycline vs Matching Placebo; The null hypothesis was that the 24 week change of fine motor/nonverbal function domain score in the minocycline group was the same as in the placebo group; Test type: Superiority or Other; p = 0.637, Regression, Linear — The p-value was not adjusted for multiple comparisons; The model was adjusted for the stratification variables, the CNS penetration score, and the baseline fine motor/nonverbal function domain score; Slope = -0.086, 95% CI 2-sided [-0.449 to 0.276], Standard Error of Mean 0.182

8. Secondary Outcome: Change in Information Processing Function Domain Z-Score
Description: The information processing function domain score is the average of age and education adjusted z scores of simple and sequential reaction time - CalCAP. The outcome is the 24 week change of information processing function domain z-scores (week 24-baseline).
Time Frame: At baseline and week 24
Population: The analysis was based on observed data.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 40 | 45
z-score | 0.14 (1.65) | 0.20 (1.14)
Statistical Analysis 1: Comparison: Minocycline vs Matching Placebo; The null hypothesis was that the 24 week change of information processing function domain score in the minocycline group was the same as the one in the placebo group; Test type: Superiority or Other; p = 0.754, Regression, Linear — The p-value was not adjusted for multiple comparisons; The model was adjusted for the stratification variables, the CNS penetration score, and the baseline information processing function domain score; Slope = -0.074, 95% CI 2-sided [-0.544 to 0.396], Standard Error of Mean 0.236

9. Secondary Outcome: Change in Verbal Memory Domain Z-Score
Description: The verbal memory domain score is the average of age and education adjusted z scores of Hopkins Verbal Learning Test- Revised, Learning and Delayed Recall. The outcome is the 24 week change of verbal memory domain z-scores (week 24-baseline).
Time Frame: At baseline and week 24
Population: The analysis was based on observed data.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 41 | 47
z-score | 0.18 (0.96) | 0.02 (1.10)
Statistical Analysis 1: Comparison: Minocycline vs Matching Placebo; The null hypothesis was that the 24 week change of verbal memory domain score in the minocycline group was the same as the one in the placebo group; Test type: Superiority or Other; p = 0.484, Regression, Linear — The p-value was not adjusted for multiple comparisons; The model was adjusted for the stratification variables, the baseline CNS penetration score, and the baseline verbal memory domain score; Slope = 0.145, 95% CI 2-sided [-0.266 to 0.558], Standard Error of Mean 0.207

10. Secondary Outcome: Change in Frontal Systems Function Domain Z-Score
Description: The frontal systems function domain score is the average of age and education adjusted z scores of Stroop Color Interference Test (CTP) and interference task (STP). The outcome is the 24 week change of frontal systems function domain z-score (week 24-baseline).
Time Frame: At baseline and week 24
Population: The analysis was based on observed data.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 41 | 47
z-score | -0.04 (0.78) | 0.21 (1.05)
Statistical Analysis 1: Comparison: Minocycline vs Matching Placebo; The null hypothesis was that the 24 week change of frontal systems function domain score in the minocycline group was the same as the one in the placebo group; Test type: Superiority or Other; p = 0.467, Regression, Linear — The p-value was not adjusted for multiple comparisons; The model was adjusted for the stratification variables, the baseline CNS penetration score, and the baseline frontal systems function domain score; Slope = -0.126, 95% CI 2-sided [-0.467 to 0.216], Standard Error of Mean 0.172

11. Secondary Outcome: Change in Karnofsky Performance Score
Description: The original Karnofsky performance score is 11 level score which ranges between 0 to 100. The score 100 means normal and 0 means death; therefore, higher score means higher ability to perform daily tasks.
  For the analysis, a new dichotomous variable (no change/worse vs. better at 24 weeks compared to baseline) was created.
Time Frame: At baseline and week 24
Population: The analysis was based on observed data.
Measure: Number; unit: participants
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 39 | 45
participants
  No Change/Worse | 33 | 42
  Better | 6 | 3
Statistical Analysis 1: Comparison: Minocycline vs Matching Placebo; The null hypothesis was that the proportion of being "better" at 24 weeks in minocycline group was the same as in the placebo group; Test type: Superiority or Other; p = 0.234, Regression, Linear — The p-value was not adjusted for multiple comparisons; The model was adjusted for the CNS penetration score. The stratification variables could not be included in the model since the model fit was poor; Odds Ratio (OR) = 2.476, 95% CI 2-sided [0.575 to 10.668], Standard Deviation 1.048

12. Secondary Outcome: Changes in Cluster of Differentiation 4 (CD4) Cell Counts (24 Weeks)
Description: The outcome was the 24 week change in CD4 cell count (week 24-baseline).
Time Frame: At baseline and weeks 24
Population: The analysis was based on observed data.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 40 | 34
cells/mm^3 | 24.10 (141.22) | 8.24 (143.02)
Statistical Analysis 1: Comparison: Minocycline vs Matching Placebo; The null hypothesis was that the 24 week change in CD4 cell counts in the minocycline group was the same as the one in the placebo group; Test type: Superiority or Other; p = 0.574, Regression, Linear — The p-value was not adjusted for multiple comparisons; The model was adjusted for stratification variables, the baseline CNS score, and the baseline CD4 cell count; Slope = 19.09, 95% CI 2-sided [-48.26 to 86.44], Standard Error of Mean 33.75

13. Secondary Outcome: Changes in Cluster of Differentiation 8 (CD8) Cell Counts (24 Weeks)
Description: The outcome was the 24 week change of CD8 cell counts (week 24-baseline).
Time Frame: At baseline and week 24
Population: The analysis was based on observed data.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 40 | 34
cells/mm^3 | 43.90 (244.51) | 0.00 (253.18)
Statistical Analysis 1: Comparison: Minocycline vs Matching Placebo; The null hypothesis was that the 24 week change in CD8 cell count in the minocycline group was the same as the one in the placebo group; Test type: Superiority or Other; p = 0.502, Regression, Linear — The p-value was not adjusted for multiple comparisons; The model was adjusted for the stratification variables, the baseline CNS penetration score, and the baseline CD8 cell counts; Slope = 40.43, 95% CI 2-sided [-79.12 to 159.97], Standard Error of Mean 59.91

14. Secondary Outcome: Number of Participants With Grade 2 or Higher Toxicity and/or Signs and Symptoms
Description: Grade or higher means that adverse events were moderate, severe, or life-threatening, or death. Grade 2 or higher adverse events are lised in the Adverse Event section.
Time Frame: Throughout study up to week 48
Population: The analysis includes all randomized participants. A total of 37 minocycline and 38 placebo participants reported Grade 2 or higher toxicity and/or signs and symptoms during 48 weeks.
Measure: Number; unit: participants with an event
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 52 | 55
participants with an event
  0 - 4 weeks | 29 | 32
  4.01 - 12 weeks | 5 | 3
  12.01 - 24 weeks | 2 | 1
  24.01 - 48 weeks | 1 | 2
Statistical Analysis 1: Comparison: Minocycline vs Matching Placebo; The null hypothesis was that the time to Grade 2 or higher toxicity and/or signs and symptoms in the minocycline group was the same as the one in the placebo group; Test type: Superiority or Other; p = 0.967, Log Rank

15. Secondary Outcome: Change of HIV Plasma RiboNucleic Acid (RNA) Viral Load
Description: The original scale of HIV RNA viral load is between 30 copies/mL to infinitive. The minimum score of 30 is the lowest detectable value. The summary table categorized this continuous value to a dichotomous variable (<30 copies/mL and >= 30 copies/mL).
Time Frame: At baseline and week 24
Population: The summary statistics were based on observed data. No statistical analysis was conducted.
Measure: Number; unit: participants
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 20 | 21
participants
  >= 30 copies/mL at base, >= 30 at week 24 | 1 | 0
  >= 30 copies/mL at base, < 30 at week 24 | 0 | 2
  < 30 copies/mL at base, >= 30 at week 24 | 2 | 0
  < 30 copies/mL at base, < 30 at week 24 | 17 | 19

16. Secondary Outcome: Changes in Instrumental Activities of Daily Living Questionnaire
Description: The Instrumental Activities of Daily Living (IADL) questionnaire is designed to learn more about how subjects are able to perform common tasks. There are 16 common tasks. For each task, if the score at the time of evaluation is worse than the best in the past, an indicator of 1 is given. Otherwise, the indicator is 0. The overall IADL score is a sum of 16 indicators divided by 16; therefore, the range is between 0 and 1 and the lower score is better. The 24-week change of IADL score was changed into a categorical variable (no change/worse vs. better) at week 24 compare to baseline.
Time Frame: At baseline and week 24
Population: The analysis was based on observed data.
Measure: Number; unit: participants
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 42 | 43
participants
  No Change/Worse | 30 | 32
  Better | 12 | 11
Statistical Analysis 1: Comparison: Minocycline vs Matching Placebo; The null hypothesis was that the proportion of participants who got better at week 24 compared to baseline in the minocycline group was the same as the one in the placebo group; Test type: Superiority or Other; p = 0.890, Regression, Logistic — The p-value was not adjusted for multiple comparisons; The model was adjusted for the stratification variables and the baseline CNS penetration score; Odds Ratio (OR) = 1.071, 95% CI 2-sided [0.405 to 2.837], Standard Error of Mean 0.497

17. Secondary Outcome: Changes in Medication Management Test (Modified)
Description: The medication management test (modified) is designed to assess participants' medication management ability and their own medications and management. It's the number of how many times participants correctly answered 16 questions. The score ranges between 0 and 16, and higher score indicates better medication management.
Time Frame: At baseline and weeks 24
Population: The analysis was based on observed data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 43 | 46
scores on a scale | 0.16 (1.57) | 0.48 (2.00)
Statistical Analysis 1: Comparison: Minocycline vs Matching Placebo; The null hypothesis was that the 24 change of medication management test score in the minocycline group was the same as the one in the placebo group; Test type: Superiority or Other; p = 0.304, Regression, Linear — The p-value was not adjusted for multiple comparisons; The model was adjusted for the stratification variables, the baseline CNS penetration score, and the baseline medication management score; Slope = -0.405, 95% CI 2-sided [-1.182 to 0.373], Standard Error of Mean 0.391

18. Secondary Outcome: Changes in Protein Markers of Oxidative Stress (Unit = Counts Per Second Only)
Description: Protein marker of oxidative stress (Ceramides, Monohexosylceramides, Dihydro Glycosyl Galceramides, and Dihexosylceramides). For all markers, the outcome is the 24 week change (week 24-baseline).
Time Frame: At pre-entry and Week 24
Population: Participants who were willing to receive the lumber punctures at week 0 and 24.
Measure: Median (Inter-Quartile Range); unit: counts per second
Arm/Group | Arm 1: Minocycline | Arm 2: Matching Placebo
Number analyzed (Participants) | 6 | 8
counts per second
  Ceramides (counts per second) | 0.0007 [-0.0001 to 0.0060] | -0.0051 [-0.0177 to 0.0006]
  Monohexosylceramides (counts per second) | 0.0013 [-0.0007 to 0.0330] | -0.0066 [-0.0279 to -0.0004]
  Dihydro Glycosyl Galceramides (counts per second) | 0.0201 [0.0043 to 0.0355] | -0.0048 [-0.0180 to -0.0010]
  Dihexosylceramides (counts per second) | 0.0005 [-0.0003 to 0.0070] | -0.0043 [-0.0090 to -0.0001]

19. Secondary Outcome: Changes in Markers of Oxidative Stress and Immune Activation (Unit=pg/mL Only)
Description: Protein markers of oxidative stress (Protein carbonyls) and markers of immune activation (TNF-a, IL-6,CXCL8, Hepatocyte growth factor, Osteopontin, sFAS, sFAS ligand, and CXCL12). For all markers, the outcome is the 24 week change (week 24-baseline).
Time Frame: At pre-entry and Week 24
Population: Participants who were willing to receive the lumber punctures at week 0 and 24.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Arm 1: Minocycline | Arm 2: Matching Placebo
Number analyzed (Participants) | 8 | 13
pg/mL
  Protein carbonyls (pg/ml) | 4.0 [3.32 to 82.29] | 13.2 [0.13 to 39.74]
  TNF-α (pg/mL) | 0.04 [0.00 to 0.31] | 0.14 [0.00 to 0.65]
  IL-6 (pg/mL) | -0.29 [-0.67 to 2.58] | 0.95 [-0.79 to 2.41]
  CXCL8 (pg/mL) | 0.34 [-3.07 to 5.97] | -6.13 [-12.5 to 3.07]
  Hepatocyte growth factor (pg/mL) | 16.09 [-21.54 to 168.99] | 90.48 [6.70 to 250.39]
  Osteopontin (pg/mL) | -5208.94 [-11579.90 to 7088.79] | 673.55 [-14689.54 to 23344.10]
  sFAS (pg/mL) | 0.68 [-9.35 to 77.79] | 134.1 [26.41 to 279.87]
  sFAS ligand (pg/mL) | -0.27 [-0.65 to 0.06] | 0.11 [-0.07 to 1.47]
  CXCL12 (pg/mL) | 204.39 [-164.20 to 1152.41] | 1,071.84 [-96.75 to 1678.84]

20. Secondary Outcome: Changes in Markers of Oxidative Stress (Unit = Pixels/mm2 Only)
Description: Protein marker of oxidative stress (Neurofilament heavy polypeptide). The outcome is the 24 week change (week 24-baseline).
Time Frame: At pre-entry and Week 24
Population: Participants who were willing to receive the lumber punctures at week 0 and 24.
Measure: Median (Inter-Quartile Range); unit: Pixels/mm^2
Arm/Group | Arm 1: Minocycline | Arm 2: Matching Placebo
Number analyzed (Participants) | 5 | 5
Pixels/mm^2 | -59.3 [-76.05 to -36.69] | -3.04 [-6.31 to 59.86]

21. Secondary Outcome: Changes in Neurotransmitter Levels (Unit = uM Only)
Description: Neurotransmitter levels (Glutamate, Tryptophan, Anthranilic Acid, Quinolinic Acid, Kynurenin, and 3-Hydroxykynurenine). The outcome is the 24 week change (week 24-baseline).
Time Frame: At pre-entry and Week 24
Population: Participants who were willing to receive the lumber punctures at week 0 and 24.
Measure: Median (Inter-Quartile Range); unit: uM
Arm/Group | Arm 1: Minocycline | Arm 2: Matching Placebo
Number analyzed (Participants) | 4 | 6
uM
  Glutamate (uM) | 5.09 [-11.01 to 13.41] | -1.08 [-1.20 to 10.88]
  Tryptophan (uM) | -0.21 [-0.78 to 0.12] | 0.07 [0.05 to 0.21]
  Anthranilic Acid (uM) | 0.0 [-2.25 to 10.87] | 0.0 [-7.14 to 6.15]
  Quinolinic Acid (uM) | -0.55 [-7.94 to 0.00] | 0.0 [-9.07 to 4.11]
  Kynurenin (uM) | 6.85 [0.01 to 46.75] | 6.97 [0.00 to 23.90]
  3-Hydroxykynurenine (uM) | -4.09 [-11.51 to 0.02] | -0.83 [-5.97 to 0.00]

22. Secondary Outcome: Changes in Alternate Psychomotor Function Z-Score
Description: The alternate psychomotor function is defined as the mean of age, sex, education, and African-American ethnicity adjusted z scores of Trail Making Part A (TMA), and age and education adjusted z score of Symbol Digit (SYD). The outcome is the 24 week change in alternate psychomotor function z-score (week 24-baseline).
Time Frame: At baseline and week 24
Population: The analysis was based on the observed data.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 41 | 48
z-score | -0.03 (0.66) | 0.05 (0.76)
Statistical Analysis 1: Comparison: Minocycline vs Matching Placebo; The null hypothesis was that the 24 week change in alternate psychomotor function score in the minocycline group was the same as the one in the placebo group; Test type: Superiority or Other; p = 0.506, Regression, Linear — The p-value was not adjusted for multiple comparisons; The model was adjusted for the stratification variables, the baseline CNS penetration score, and the baseline alternate psychomotor function score; Slope = -0.097, 95% CI 2-sided [-0.388 to 0.193], Standard Error of Mean 0.146

23. Secondary Outcome: Changes in Alternate Verbal Memory Z-Score
Description: The alternate verbal memory was defined as a mean of age and education adjusted z score of trials 1 to 3 and delayed recall tests. The outcome is the 24 week change in alternate verbal memory z-score (week 24-baseline).
Time Frame: At baseline and week 24
Population: The analysis is based on observed data.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 41 | 47
z-score | 0.18 (0.96) | 0.02 (1.10)
Statistical Analysis 1: Comparison: Minocycline vs Matching Placebo; The null hypothesis was that the 24 week change in the alternate verbal memory score in the minocycline group was the same as the one in the placebo group; Test type: Superiority or Other; p = 0.484, Regression, Linear — The p-value was not adjusted for multiple comparisons; The model was adjusted for stratification variables, baseline CNS penetration score, and the baseline alternate verbal memory score; Slope = 0.146, 95% CI 2-sided [-0.266 to 0.558], Standard Error of Mean 0.207

24. Secondary Outcome: Changes in Alternate Frontal Systems Z-Score
Description: The alternate frontal systems was defined as a mean of age and education adjusted z score of Interference task, and age, sex, education, and African-American ethnicity adjusted z score of Trail Making Part B. The outcome was the 24 week change in alternate frontal systems z-score (week 24-baseline).
Time Frame: At baseline and week 24
Population: The analysis was based on observed data.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Minocycline | Matching Placebo
Number analyzed (Participants) | 41 | 47
z-score | 0.03 (0.67) | -0.07 (0.70)
Statistical Analysis 1: Comparison: Minocycline vs Matching Placebo; The null hypothesis was the 24 week change of alternate frontal systems score in the minocycline group was the same as the one in the placebo group; Test type: Superiority or Other; p = 0.690, Regression, Linear — The p-value was not adjusted for multiple comparisons; The model was adjusted for stratification variables, baseline CNS penetration score, and the baseline alternate frontal systems score; Slope = 0.055, 95% CI 2-sided [-0.217 to 0.327], Standard Error of Mean 0.137

ADVERSE EVENTS:
Time Frame: Up to 48 weeks since the randomization.
Arm/Group | Minocycline | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 7/52 | 3/55
Other Adverse Events (participants affected / at risk) | 18/52 | 34/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (N=52) | Matching Placebo (N=55)
Blood amylase increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Grade 4: Life-threatening
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0) — Amyotrophic lateral sclerosis (ALS)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) — Requires dialysis
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — On nose
Tooth infection (General disorders) | 1 (1) | 0 (0) — Tooth discoloration
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) — Resulted in hospitalization
Suicidal attempt (Psychiatric disorders) | 0 (0) | 1 (1) — By medication overdose
Hypertension (General disorders) | 0 (0) | 1 (1)
Blood triglycerides increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (N=52) | Matching Placebo (N=55)
Fatigue (General disorders) | 4 (4) | 3 (3)
Pain (General disorders) | 5 (9) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Sob (General disorders) | 0 (0) | 4 (4)
Diarrhea/Loose (Gastrointestinal disorders) | 5 (5) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4)
Headache (General disorders) | 1 (1) | 7 (7)

LIMITATIONS AND CAVEATS:
Originally, 100 participants were expected to enroll. As of the early termination notice, 107 participants were randomized, yet not all subjects could complete the 24 week assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trial Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.